CLINICAL TRIAL: NCT05873686
Title: A Phase 1 Clinical Study of NXP900 in Subjects With Advanced Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvectis Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NXP900-101
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor; NSCLC (Non-small Cell Lung Cancer); Renal Cancer; Mesothelioma; Non-Small Cell Squamous Lung Cancer; Non-small Cell Lung Adenocarcinoma
Keywords: Solid Tumor; Carcinoma; Neoplasms; Adenocarcinoma; YES1; YAP1; TAZ1; NF2; FAT1; LATS1; TYMS; gene amplification; gene mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Kidney Neoplasms; Mesothelioma; Carcinoma; Neoplasms; Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Sequential assignment, dose escalation and expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Part A) (Experimental): Escalating doses of NXP900 are planned with a starting dose level of 20 mg once per day.
  Interventions: Drug: NXP900
- Dose Expansion (Part B) (Experimental): Participants will receive the selected dose of NXP900
  Interventions: Drug: NXP900

INTERVENTIONS:
Drug: NXP900 — NXP900 is an orally administered SRC/YES1 kinase inhibitor

SUMMARY:
This is a multi-center, first-in-human, open label, dose escalation (Part A) and expansion (Part B) Phase 1 study in subjects with advanced solid tumors and in subjects with solid tumors with selected genetic alterations that are either direct (YES1 amplification) or dependent (Hippo Pathway alterations) targets of NXP900.

ELIGIBILITY:
Part A

Inclusion Criteria:

1. Provide written informed consent.
2. 18 years old or older.
3. Advanced, metastatic, and/or progressive solid tumors for whom there is no authorized or effective therapy available, or for whom such therapies are considered inappropriate by the Investigator.
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

1. Subjects with known human epidermal growth factor receptor 2 (HER2+) overexpressing malignancies.
2. Radiotherapy (except for palliative reasons), endocrine therapy, chemotherapy, or investigational agent within 28 days, (42 days for nitrosoureas, mitomycin-C) of first dose of NXP900. Subjects can continue to receive bisphosphonates due to metastatic bone disease or GnRH agonists if they have prostate cancer.
3. Ongoing toxic manifestations of previous treatments > Grade 2 with the exception of alopecia and neuropathy.
4. Subjects with treated brain metastases with evidence of progression within 28 days after central nervous system (CNS)-directed treatment, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan) during the Screening period.
5. Female subjects who can become pregnant (or are already pregnant or lactating), unless they have a negative serum pregnancy test before enrollment and agree to use at least one highly effective form of contraception .
6. Male subjects with partners of childbearing potential, unless they agree to take measures not to father children by using a barrier method of contraception (condom plus spermicide).
7. Major surgery from which the subject has not yet recovered.

Part B:

Inclusion Criteria:

1. Provide written informed consent.
2. 18 years old or older.
3. Advanced, metastatic, and/or progressive solid tumors with pathogenic molecular alterations:

   1. Non-small cell lung cancer (adenocarcinoma); YES1, TYMS amplification or FAT1 pathogenic mutation
   2. Non-small cell lung cancer (squamous cell carcinoma); YES1, TYMS amplification or FAT1 pathogenic mutation
   3. Renal cancer; NF2 pathogenic mutation
   4. Mesothelioma; NF2 pathogenic mutation
   5. Other solid tumors with a NF2, FAT1 or LATS1 pathogenic gene mutation or TYMS, YAP1, YES1, TAZ1 gene amplification
4. Must have received 1-3 prior therapies appropriate for their tumor type and stage of disease
5. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

1. Subjects with the following combination of cancer type and pathogenic molecular alterations are excluded:

   1. Subjects with colorectal cancer, glioma, melanoma, or anaplastic thyroid conditions with BRAF mutations.
   2. Subjects with NSCLC with BRAF, EGFR or HER2 alterations.
   3. Subjects with breast cancer, gastric cancer, esophageal junction adenocarcinoma or biliary cancer with HER2 alterations,
2. Subjects with anal, penile, cervical or head and neck cancers with a prior history of human papilloma virus (HPV) infection.
3. Radiotherapy (except for palliative reasons), endocrine therapy, chemotherapy, or investigational agent within 28 days (42 days for nitrosoureas, mitomycin-C) prior to first dose of NXP900. Subjects can continue to receive bisphosphonates due to metastatic bone disease or GnRH agonists if they have prostate cancer.
4. Ongoing toxic manifestations of previous treatments > Grade 2 with the exception of alopecia and neuropathy.
5. Female subjects who can become pregnant (or are already pregnant or lactating), unless they have a negative serum pregnancy test before enrollment and agree to use at least one highly effective form of contraception .
6. Male subjects with partners of childbearing potential, unless they agree to take measures not to father children by using a barrier method of contraception (condom plus spermicide).
7. Major surgery from which the subject has not yet recovered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment related adverse events and/or clinical laboratory abnormalities | Up to 30 days post treatment
Part A: Number of patients who experience Dose Limiting Toxicities (DLT) as defined in the protocol | Day 28
Part B: Objective response rate (ORR) | Up to 24 months
  Best response of complete response (CR) or partial response (PR) per RECIST 1.1
Part B: Duration of Response (DoR) | Up to 24 months
  Confirmed CR or PR from the first documented response to the date of documented disease progression or death.
Part B: Disease Control Rate (DCR) | Up to 24 months
  The proportion of patients with stable disease (SD), partial response (PR), or complete response (CR).

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) of NXP900 | Up to 24 months
Maximum observed concentration (Cmax) of NXP900 | Up to 24 months
Time to peak concentration (Tmax) of NXP900 | Up to 24 months
Half-life (T1/2) of NXP900 | Up to 24 months
Apparent volume of distribution at steady state (Vss/F) of NXP900 | Up to 24 months
Apparent plasma clearance at steady state (Clss/F) of NXP900 | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Udai Banerji, Prof, Principal Investigator — Institute of Cancer Research, Royal Marsden NHS Foundation Trust; Gerald Falchook, MD, Principal Investigator — Sarah Cannon Cancer Institute, HealthOne Denver
Locations (7):
- United States (5):
  - Mayo Clinic, Phoenix, Arizona
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Oregon Health and Science University, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- United Kingdom (2):
  - Western General Hospital - NHS Lothian, Edinburgh
  - The Royal Marsden NHS Foundation and Trust, London

IPD SHARING:
Plan to Share IPD: No